CLINICAL TRIAL: NCT03321279
Title: Social Incentives to Increase Mobility Among Hospitalized Patients: The MOVE IT Randomized Trial
Brief Title: Social Incentives to Increase Mobility
Acronym: MOVE IT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 826974
Record Dates: First submitted 2017-10-04; First posted 2017-10-25 (Actual); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Pneumonia; Diabetes; Congestive Heart Failure; Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pneumonia; Diabetes Mellitus; Heart Failure; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Participants' daily step counts will be for weeks 2-13 after hospital discharge. Participants will be asked to complete surveys at 5, 9 and 13 weeks post-discharge.
- Intervention (Experimental): Participants' daily step counts will be monitored for weeks 2-13 after hospital discharge. Participants will have a weekly step goal that increases from baseline by 10% each week of the intervention (12 weeks). Participants will engage in a social incentive-based gamification based on points and levels that leverages loss aversion, which has been demonstrated to motivate behavior change more effectively with losses than gains. Participants will receive daily feedback for the step counts and weekly feedback for levels. Participants will be asked to identify a support partner, who will receive weekly reports with the the participant's points and levels balance.
  Interventions: Behavioral: Social Incentive

INTERVENTIONS:
Behavioral: Social Incentive — Participants in the intervention arm will receive social incentives as part of the intervention. See arm descriptions for more detail.
  Arms: Intervention

SUMMARY:
This study aims to assess the effectiveness of a social incentive-based gamification intervention to increase physical activity in the 3 months after hospital discharge.

DETAILED DESCRIPTION:
This study aims to assess the effectiveness of a social incentive-based gamification intervention to increase physical activity in the 3 months after hospital discharge. To do this, the investigators will conduct a two-arm randomized, controlled trial during the 3-months after hospital discharge comparing a control group that uses a wearable device to track physical activity to an intervention group that uses the same wearable devices and receives a supportive social incentive-based gamification intervention to adhere to a step goal program. Patients will be enrolled during hospitalization from medicine and oncology floors into three phases. In phase 1 (hospitalization), patients inpatient step counts will be monitored. In phase 2 (week 1 post-discharge), patients will have a baseline step count estimated. In phase 3 (weeks 2-13 post-discharge), patients will be randomly assigned to the control or intervention group. Patients will be considered enrolled in the trial if they complete the run-in periods (phases 1 and 2) and then are randomized into phase 3.

The enrollment phase will be part of another randomized trial which evaluates the impact of three recruitment strategies on patient enrollment. This trial will be completed and unmasked to patients before they begin the phase 1 of our study.

The investigators will also explore patients' physical activity while in the hospital and if that differs across floors that have or have not deployed a nursing mobility protocol. Changes in patient functional decline and 30-day hospital readmission will also be explored.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Admitted to medicine or oncology floor in the hospital

Exclusion Criteria:

* Inability to provide informed consent
* Does not have daily access to a smartphone compatible with the wearable device
* Already enrolled in another physical activity program
* Inpatient mobility score of 0 or 1 indicating that physical activity is not appropriate for the patient
* Any other medical conditions that would prohibit participation in a 3-month physical activity program
* Unable to complete the run-in phases (e.g. not discharged from the hospital within 60 days of enrolling; not willing to use the wearable device for the 3-month post-discharge intervention).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 233 (Actual)
Dates: Start 2018-01-11 (Actual); Primary Completion 2019-09-09 (Actual); Study Completion 2019-09-09 (Actual)

PRIMARY OUTCOMES:
Change in mean daily step count from the baseline period to the intervention period, using a wearable pedometer (Nokia Steel) to measure step count. | 13 weeks
  The primary outcome variable is the change in mean daily step count from the baseline period (week 1 post-discharge) to the intervention period (weeks 2-13 post-discharge). This will be measured using the Nokia Steel wearable device. .

SECONDARY OUTCOMES:
30-day hospital readmission post-discharge, using the state's hospital database | 13 weeks
  A secondary outcome variable is 30-day hospital readmission post-discharge, which will be obtained from the state-based registry.
Functional decline from admission to 3 months post-discharge, measured using validated survey assessments. | 13 weeks
  A secondary outcome variable is functional decline from admission to 3 months post-discharge, which will be obtained from information collected through validated survey assessments.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Greysen, MD, MHS, MA, Principal Investigator — University of Pennsylvania; Mitesh Patel, MD, MBA, MS, Study Director — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Willinger CM, Waddell KJ, Arora V, Patel MS, Ryan Greysen S. Patient-reported sleep and physical function during and after hospitalization. Sleep Health. 2024 Apr;10(2):249-254. doi: 10.1016/j.sleh.2023.12.001. Epub 2023 Dec 26. PMID 38151376
- [Derived] Greysen SR, Waddell KJ, Patel MS. Exploring Wearables to Focus on the "Sweet Spot" of Physical Activity and Sleep After Hospitalization: Secondary Analysis. JMIR Mhealth Uhealth. 2022 Apr 27;10(4):e30089. doi: 10.2196/30089. PMID 35476034
- [Derived] Greysen SR, Changolkar S, Small DS, Reale C, Rareshide CAL, Mercede A, Snider CK, Greysen HM, Trotta R, Halpern SD, Patel MS. Effect of Behaviorally Designed Gamification With a Social Support Partner to Increase Mobility After Hospital Discharge: A Randomized Clinical Trial. JAMA Netw Open. 2021 Mar 1;4(3):e210952. doi: 10.1001/jamanetworkopen.2021.0952. PMID 33760089
- [Derived] Greysen HM, Reale C, Mercede A, Patel MS, Small D, Snider C, Rareshide C, Halpern SD, Greysen SR. Mobility and outcomes for validated evidence - Incentive trial (MOVE IT): Randomized clinical trial study protocol. Contemp Clin Trials. 2020 Feb;89:105911. doi: 10.1016/j.cct.2019.105911. Epub 2019 Dec 12. No abstract available. PMID 31838257